CLINICAL TRIAL: NCT06928922
Title: The Phase I Clinical Study of the Inhaled mRNA Tumor-associated Antigen Dry Powder Vaccine BMD006 in Patients With Advanced Lung Cancer or Metastatic Solid Tumors in the Lungs.
Brief Title: Inhaled mRNA Tumor-associated Antigen Dry Powder Vaccine in Advanced Lung Cancer and Lung Metastasis of Solid Tumors.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BMD006-001
Record Dates: First submitted 2025-03-26; First posted 2025-04-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Advanced Lung Cancer; Lung Metastasis
Keywords: inhaled mRNA tumor-associated antigen dry powder vaccine; advanced lung cancer; solid tumors with lung metastasis; mRNA vaccine combination with PD-1 or PD-1/VEGF antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BMD006 monotreatment (Experimental): BMD006 is packaged in capsules and contains white powder. Under no circumstances should it be swallowed, and only the Breezhaler inhalation device (consisting of a dust cap, nozzle, base, puncture button, and central chamber) should be used for inhalation therapy.
  BMD006 monotreatment is treated on D1, D15, and D22, and D28 is evaluated by investigators to be safe and tolerable. The patient will continue to receive QW treatment at the current dose level for 6 times, and then switch to Q3W treatment until 52 weeks after the first treatment or reaching the termination criteria.
  Interventions: Biological: BMD006 monotreatment
- BMD006 in combination with PD-1or PD-1/VEGF antibody (Experimental): BMD006 was treated at D1, D8, and D15, and D21 was evaluated by researchers to be safe and tolerable. The patient will continue to receive QW treatment at the current dose level for 6 times, and then switch to Q3W treatment until 52 weeks after the first treatment or until the termination criteria are met in BMD006 in combination with PD-1 or PD-1/VEGF antibody.
  PD-1 antibodies will be used according to medical advice and instructions.
  Interventions: Biological: BMD006 in combination with PD-1 antibody
- BMD006 in combination with PD-1/VEGF antibody (Experimental): The subjects will be randomly assigned in a 1:1 ratio to either the BMD006 and PD-1/VEGF group (Group 1) or the BMD006 monotherapy group for six weeks plus two drugs combination therapy group (Group 2). The ratio of the two groups will be 1:1, with no less than 10 patients in each group.
  The first group is a combination therapy of BMD006 and PD-1/VEGF. BMD006 is administered once a week for the first six weeks, and will be adjusted to once every three weeks starting from the seventh week. PD-1/VEGF is administered once every three weeks. The second group received BMD006 monotherapy once a week, and after six doses, the researchers evaluated the potential benefits. Starting from the seventh week, BMD006 was used in combination with PD-1/VEGF, and thereafter BMD006 was used every three weeks, while PD-1/VEGF was used every three weeks.
  Interventions: Biological: BMD006 in combination with PD-1/VEGF antibody

INTERVENTIONS:
Biological: BMD006 monotreatment — After receiving the first dose of BMD006 treatment on Day 1, the patient will complete a single-treatment DLT observation (14 days). If the treatment is deemed safe and tolerable by the investigator, the patient will proceed to multiple-treatment DLT observation (14 days), with BMD006 treatment administered on Day 15 and Day 22. On Day 28, if the treatment is again assessed as safe and tolerable by the investigator, the patient will continue treatment at the current dose level following a QW (once weekly) regimen for 6 doses. After that, starting from Week 11, the treatment schedule will change to Q3W (once every 3 weeks) until 52 weeks after the first treatment or until the treatment discontinuation criteria are met.
  Arms: BMD006 monotreatment
Biological: BMD006 in combination with PD-1 antibody — Once the dose escalation of BMD006 monotreatment is completed and the MTD (Maximum Tolerated Dose) is determined (i.e., the RP2D for this study), a dose escalation exploration of BMD006 in combination with PD-1 antibody will be conducted. On Day 1, patients will receive BMD006 in combination with PD-1 antibody treatment, followed by BMD006 treatment on Days 8 and 15. The DLT observation period will be 21 days. On Day 21, if the treatment is assessed as safe and tolerable by the investigator, the patient will continue treatment at the current dose level according to the QW (once weekly) regimen for 6 doses. After Week 10, the treatment schedule will change to Q3W (once every 3 weeks) until 52 weeks after the first treatment or until the treatment discontinuation criteria are met.
  Arms: BMD006 in combination with PD-1or PD-1/VEGF antibody
Biological: BMD006 in combination with PD-1/VEGF antibody — The first group is a combination therapy of BMD006 and PD-1/VEGF. BMD006 was administered once a week for the first six weeks, and adjusted to once every three weeks starting from the seventh week. PD-1/VEGF was administered once every three weeks. The second group received BMD006 monotherapy once a week. After six doses, the researchers evaluated the potential benefits and started using PD-1/VEGF in combination from the seventh week onwards. BMD006 was then administered every three weeks, and PD-1/VEGF was administered every three weeks thereafter
  Arms: BMD006 in combination with PD-1/VEGF antibody

SUMMARY:
BMD006 is an inhaled mRNA tumor-associated antigen dry powder vaccine targeting lung cancer and solid tumors with lung metastasis, classified as an off-the-shelf anti-tumor product. The product contains two clinically validated TAA antigen combinations: for patients with solid tumors that have lung metastasis, the mRNA vaccine consists of four mRNA sequences encoding melanoma-associated tumor antigens ; for patients with primary lung cancer, the mRNA vaccine consists of six mRNA sequences encoding tumor-associated antigens of primary lung cancer .

This study is a single-center, open-label, dose-escalation trial designed to evaluate the safety, tolerability, preliminary efficacy, PK, and PD of BMD006 in patients with advanced lung cancer or advanced solid tumors with lung metastasis who have failed standard treatments or have no standard treatment options. Additionally, the study will further explore the effect of BMD006 in combination with PD-1 or Ivonescimab Injection treatment.

DETAILED DESCRIPTION:
This study adopts a single center, open label, dose escalation design to evaluate the safety, tolerability, preliminary efficacy, PK and PD characteristics of BMD006 in patients with advanced lung cancer or advanced solid tumors with lung metastasis who have failed standard treatment or have no standard treatment, and to explore the treatment of BMD006 PD-1 or PD-1/VEGF.

This study includes three parts: exploring the dosage of BMD006 alone, exploring the dosage of BMD006 combined with PD-1 or PD-1/VEGF, and expanding the dosage of BMD006 combined with PD-1/VEGF.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with the requirements of the study protocol, voluntarily participate in the trial, and sign a written informed consent form (ICF).
* Must be at least 18 (inclusive) at the time of signing the ICF, and both male and female participants are eligible.
* Histologically or cytologically confirmed as advanced lung cancer (driver gene negative) or advanced solid tumors with lung metastasis, and having failed prior standard treatments or having no standard treatment options.
* Agree to provide fresh tumor tissue samples or archived tumor tissue samples within the past three years.
* Presence of at least one measurable lesion as defined by RECIST V1.1
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1
* Organ function must be adequate at screening (no need for blood transfusion, hematopoietic growth factors, human albumin, or medications for correction within 14 days prior to first treatment), specifically defined as: a) Hematology: Absolute neutrophil count ≥1.5×10^9/L; platelet count ≥90×10^9/L; hemoglobin ≥90 g/L (9 g/dL). b) Liver Function: Serum total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN); for patients with liver metastasis or a history/suspected history of Gilbert's syndrome (persistent or recurrent hyperbilirubinemia, primarily unconjugated bilirubin, with no evidence of hemolysis or liver pathology), TBIL ≤3×ULN; for patients without liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST); for patients with liver metastasis, ALT or AST ≤5×ULN. c) Renal Function: Creatinine (Cr) ≤1.5×ULN or creatinine clearance (CLcr) ≥60 mL/min (calculated using the Cockcroft-Gault formula, see Attachment 3); urine dipstick test result showing urinary protein <2+; for patients with baseline urine dipstick showing protein ≥2+, a 24-hour urine collection should be conducted, and the protein content in the 24-hour urine should be <1 g. d) Cardiac Function: Echocardiography showing left ventricular ejection fraction (LVEF) >50%. e) Pulmonary Function: Shortness of breath ≤Grade 1 as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), and outdoor ambient air oxygen saturation (SpO₂) ≥92%.
* Expected life expectancy ≥12 weeks.
* Female patients of childbearing potential and male patients (and their female partners) must use highly effective contraception from the screening period until at least 6 months after the last dose of the study drug. Patients must not plan to conceive, donate sperm, or donate eggs during this period

Exclusion Criteria:

* Patients with lung cancer who have concurrent other types of malignant tumors or are diagnosed with multiple primary malignancies, except for the following: completely resected basal cell carcinoma and squamous cell carcinoma of the skin, completely resected any type of carcinoma in situ.
* Symptomatic central nervous system metastasis; for patients with asymptomatic brain metastasis or those whose symptoms have been stable for ≥2 weeks after treatment of brain metastasis, they may participate in this study if they meet all the following criteria: measurable lesions in the lungs; cessation of steroid treatment 14 days prior to the first trial product dose.
* Patients with chronic obstructive pulmonary disease (COPD), asthma, or allergies to pollen or dust.
* Patients suspected of having active or latent tuberculosis infection, based on interferon-γ release assay results, clinical symptoms, and/or chest imaging findings (patients with evidence of adequately treated prior active tuberculosis infection may be enrolled after assessment by the investigator; for latent tuberculosis, patients must have completed at least 4 weeks of anti-tuberculosis treatment, with no liver function impairment [ALT ≤3×ULN, AST ≤3×ULN], and after the investigator assesses that the risk is manageable, they may be considered for continued screening or enrollment).
* History of interstitial lung disease (e.g., idiopathic pulmonary fibrosis or organizing pneumonia), or active, non-infectious pneumonia requiring immunosuppressive treatment such as corticosteroids.
* Patients with active autoimmune diseases requiring therapeutic intervention.
* History of serious bleeding disorders; or those with coagulation dysfunction (as indicated by laboratory tests or medical history) who are deemed by the investigator to be unsuitable for the trial treatment.
* History or current diagnosis of cardiovascular disease, including any of the following: a) Recent myocardial infarction or coronary artery bypass grafting (CABG) within the past 6 months; b) Uncontrolled congestive heart failure; c) Unstable angina (within the past 6 months); d) Clinically significant (symptomatic) arrhythmias (e.g., sustained ventricular tachycardia, clinically significant second- or third-degree atrioventricular block without a pacemaker).
* Clinically uncontrolled third-space fluid accumulation (e.g., pleural effusion/pericardial effusion; patients with effusions that do not require drainage or those whose effusions have not increased significantly after stopping drainage for 3 days may be included).
* Severe infection requiring intravenous antibiotic treatment or hospitalization at screening, or any uncontrolled active infection within 4 weeks prior to the first dose of the trial product.
* History of severe allergic reactions, or known allergy to any active or inactive component of BMD006 or PD-1 inhibitors.
* Any other metabolic, hematological, renal, hepatic, pulmonary, neurological, endocrine, cardiac, or gastrointestinal disease that, in the investigator's opinion, may present unacceptable risks to the patient during treatment.
* Presence of unresolved toxicity from prior anti-tumor treatments before the first dose of the study product, which has not recovered to Grade 0 or 1 (excluding alopecia) (severity assessed according to NCI CTCAE v5.0).
* Positive test results for hepatitis B at screening [defined as: ① Hepatitis B surface antigen (HBsAg) positive; ② HBsAg negative but hepatitis B core antibody (HbcAb) positive (further testing through hepatitis B virus deoxyribonucleic acid [HBV DNA] is required, and patients with HBV DNA levels exceeding the normal limit for the test method must be excluded)], positive hepatitis C antibody (HCV Ab) [further testing through hepatitis C virus ribonucleic acid (HCV RNA) is required, and patients with HCV RNA levels exceeding the normal limit for the test method must be excluded], or positive human immunodeficiency virus antibody (HIV Ab).
* Underwent major surgery within 4 weeks prior to the first dose of the trial product (cranial, thoracic, or abdominal surgery) or has an unresolved wound, ulcer, or fracture. Note: Thoracoscopic surgery and mediastinoscopy will not be considered major surgery. Patients who are ≥2 weeks post-surgery or who are deemed eligible by the investigator may be included in the study.
* Previously received similar products or treatments.
* Received other anti-tumor treatments (radiotherapy, chemotherapy, endocrine therapy, targeted therapy, immunotherapy, etc.) within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose of the trial product.
* Received systemic immunosuppressive agents (e.g., systemic corticosteroids) within 3 months prior to the first dose of the trial product.
* Received or planned to receive live or attenuated live vaccines within 3 months prior to the first dose of the trial product or during the study.
* Pregnant or breastfeeding women.
* Participated in any clinical drug trial (defined as being randomized and receiving trial product treatment) within 3 months or 5 half-lives (whichever is longer) prior to screening.
* Any other condition deemed by the investigator to make the patient unsuitable for participation in the trial.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-02-24 (Estimated); Study Completion 2028-02-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities（DLTs） | about 2 years
  Number of participants experiencing dose-limiting toxicities（DLTs）
Determine the maximum tolerated dose（MTD） of BMD006 | about 2 years
  Determine the maximum tolerated dose（MTD） of BMD006
Determine the recommended phase II dose (RP2D) for the clinical study. | about 2 years
  Determine the recommended phase II dose (RP2D) for the clinical study.
number of participants experiencing adverse events（AEs） | about 2 years
  number of participants experiencing adverse events（AEs）

SECONDARY OUTCOMES:
overall response rate（ORR） | Up to 12 months
  The percentage of patients who achieved the best overall response of complete response (CR) or partial response (PR) as evaluated by investigators based on RECIST V1.1
Disease Control Rate(DCR) | Up to 12 months
  The percentage of patients who achieved CR, PR, or SD)as assessed by investigators based on RECIST V1.1.
Duration of Response(DOR) | Up to 12 months
  The investigators evaluated the time from objective remission to the first recorded disease progression or death (whichever occurred first) based on RECIST V1.1;
Progression-Free Survival (PFS) | Up to 12 months
  The time between the first treatment date and the date of the first recorded disease progression or death (whichever occurs first) evaluated by the investigator according to RECIST V1.1;
Overall Survival(OS) | Up to 12 months
  The time between the first treatment date and the date of the patient's death due to any reason.
The 6-month and 12-month overall survival (OS) rates. | Up to 6 or 12 months
  The 6-month and 12-month overall survival (OS) rates.
The proportion and activation status of antigen-specific T cells in peripheral blood and tumor tissue (if available) | about 2 years
  The proportion and activation status of antigen-specific T cells in peripheral blood and tumor tissue (if available)
The titers of antigen-specific antibodies IgG and IgA in serum | about 2 years
  The titers of antigen-specific antibodies IgG and IgA in serum

OTHER OUTCOMES:
Copy number of BMD006 mRNA in serum | about 2 years
  Copy number of BMD006 mRNA in serum
Circulating tumor DNA (ctDNA) levels in patients with advanced lung cancer or advanced solid tumors with lung metastasis. | about 2 years
  Circulating tumor DNA (ctDNA) levels in patients with advanced lung cancer or advanced solid tumors with lung metastasis.
The incidence of dose-limiting toxicity (DLT) after treatment with BMD006 in combination with PD-1 antibody | about 2 years
  The incidence of dose-limiting toxicity (DLT) after treatment with BMD006 in combination with PD-1 antibody
The incidence of Adverse Events (AEs) after treatment with BMD006 in combination with PD-1 antibody | about 2 years
  The incidence of Adverse Events (AEs) after treatment with BMD006 in combination with PD-1 antibody
The proportion and activation status of antigen-specific T cells in peripheral blood and tumor tissue (if available) after treatment with BMD006 in combination with PD-1 antibody | about 2 years
  The proportion and activation status of antigen-specific T cells in peripheral blood and tumor tissue (if available) after treatment with BMD006 in combination with PD-1 antibody
The titers of antigen-specific antibodies IgG and IgA in serum after treatment with BMD006 in combination with PD-1 antibody | about 2 years
  The titers of antigen-specific antibodies IgG and IgA in serum after treatment with BMD006 in combination with PD-1 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China